CLINICAL TRIAL: NCT04237727
Title: CAvent-Ventilation During Advanced Cardiopulmonary Resuscitation in Out-of-hospital Cardiac Arrest- a Descriptive Study
Acronym: CAvent
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Collaborators: Regionale Ambulance Voorziening, Amersfoort, Utrecht, Netherlands (Unknown)
Responsible Party: Principal Investigator, Sten Rubertsson, Professor, Uppsala University
Other Study IDs: VENT001
Record Dates: First submitted 2019-04-04; First posted 2020-01-23 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Out-of-Hospital Cardiac Arrest; Pulmonary Ventilation
Keywords: Out-of-Hospital Cardiac Arrest; Cardiopulmonary Resuscitation; Respiration, Artificial
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fluxmed GrH will be used to measure the ventilation parameters — The study will be a prospective descriptive multicenter study where measurement of ventilation data will be sampled during CPR by EMS treating patients with OHCA.

SUMMARY:
The aim with this descriptive multicenter study is to examine the quality of the ventilation given by Emergency Medical Service (EMS) personnel during cardiopulmonary resuscitation (CPR).

Primary endpoint is the ventilation quality measured as ventilation frequency, tidal volume and minute ventilation.

This will primarily be studied during CPR with a 30 compression/2 ventilation ratio performed by the EMS personnel where the airway is managed with a supraglottic device but also in CPR with continuous ventilation (8-10 breaths/minute) after the airway management have been replaced with an endotracheal within the emergency room.

The inclusion of patients will be performed at two sites (Uppsala; Sweden and Utrecht; Holland), all out-of-hospital cardia arrest (OHCA) patients will receive care according to current CPR guidelines using mechanical chest compressions.

DETAILED DESCRIPTION:
The inclusion is estimated to run over a two-year period to reach the goal of at least 200 patients. The study has been preceded by a trial period in an effort to solve any logistic and technical problems.

The study will be a prospective descriptive multicenter study where measurement of ventilation data will be sampled during CPR by EMS treating patients with OHCA. Any results from standard laboratory tests related to ventilation quality will be retracted from the patient medical journal systems. In addition to ventilatory variables measured as endpoints, secondary endpoints will also be outcome measures as any ROSC, survival and neurological outcome (mRS, GOS-E) measured at 30 days and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

Out-of-hospital cardiac arrest (OHCA) treated with CPR performed by the EMS personnel

Exclusion Criteria:

* Patient age < 18 years
* Known pregnancy
* Trauma related cardiac arrest (inc. hanging)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population will be patients who have suffered an OHCA with CPR started by EMS personnel in Uppsala; Sweden and Utrech, Amersfoort; Holland.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-03-29 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Ventilation frequency | From start of CPR to end of CPR.
  Measured as ventilations per minute.
Tidal volume | From start of CPR to end of CPR.
  Measured as milliliters per ventilation.
Minute Ventilation | From start of CPR to end of CPR.
  Measured as litres per minute.

SECONDARY OUTCOMES:
Variation of etCO2 in relation to different ratios of compression to ventilations | From start of CPR to end of CPR.
  etCO2 measured as kilopascal for each exhalation during CPR with 30 compressions and 2 ventilations and during continous compressions and ventilations.
Time of inspiration | From start to end of CPR.
  Measured as seconds for each inspiration.
Fraction of dead space ventilation | From start of CPR to end of CPR..
  Dead space measured as milliliters for each ventilation compared to the tidal volume in milliters for that same ventilation.
Peak inspiratory pressure during ventilation | From start of CPR to end of CPR.
  Measured as cmH20 for each ventilation.
Survival rate | 30 days post cardiac arrest
  Number of patients that has survived after the cardiac arrest.
Neurological outcome | 30 days post cardiac arrest
  Measured with the modified Ranking Scale (mRS).
Neurological outcome | 30 days post cardiac arrest.
  Measured with the Glascow Outcome Scale -Extended (GOS-E).
Survival rate | 6 months post cardiac arrest
  Number of patients that has survived after the cardiac arrest..
Neurological outcome | 6 months post cardiac arrest
  Measured with the modified Ranking Scale (mRS).
Neurological outcome | 6 months post cardiac arrest.
  Measured with the Glascow Outcome Scale -Extended (GOS-E).

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rubertsson, PhD, Principal Investigator — Uppsala University department of surgical sciences; David Smekal, PhD, Study Chair — Uppsala University department of surgical sciences; Johan Mällberg, BsSC, Study Chair — Uppsala University department of surgical sciences; René Boomars, MSc, Study Chair — Regionale Ambulance Voorziening Utrecht (RAVU); Thijs Verhagen, MD, Study Chair — Regionale Ambulance Voorziening Utrecht (RAVU)
Locations (2):
- Regionale Ambulance Voorziening Utrecht, Netherlands, Amersfoort, Utrecht, Netherlands
- Uppsala University hospital, Uppsala, Sweden

REFERENCES:
- [Background] Perkins GD, Handley AJ, Koster RW, Castren M, Smyth MA, Olasveengen T, Monsieurs KG, Raffay V, Grasner JT, Wenzel V, Ristagno G, Soar J; Adult basic life support and automated external defibrillation section Collaborators. European Resuscitation Council Guidelines for Resuscitation 2015: Section 2. Adult basic life support and automated external defibrillation. Resuscitation. 2015 Oct;95:81-99. doi: 10.1016/j.resuscitation.2015.07.015. Epub 2015 Oct 15. No abstract available. PMID 26477420
- [Background] Nizhenkovska IV, Pidchenko VT, Bychkova NG, Bisko NA, Rodnichenko AY, Kozyko NO. Influence of Ganoderma lucidum (Curt.: Fr.) P. Karst. on T-cell-mediated immunity in normal and immunosuppressed mice line CBA/Ca. Ceska Slov Farm. 2015 Sep;64(4):139-43. PMID 26459128
- [Background] Hollenberg J, Svensson L, Rosenqvist M. Out-of-hospital cardiac arrest: 10 years of progress in research and treatment. J Intern Med. 2013 Jun;273(6):572-83. doi: 10.1111/joim.12064. Epub 2013 Apr 1. PMID 23480824
- [Background] Grasner JT, Lefering R, Koster RW, Masterson S, Bottiger BW, Herlitz J, Wnent J, Tjelmeland IB, Ortiz FR, Maurer H, Baubin M, Mols P, Hadzibegovic I, Ioannides M, Skulec R, Wissenberg M, Salo A, Hubert H, Nikolaou NI, Loczi G, Svavarsdottir H, Semeraro F, Wright PJ, Clarens C, Pijls R, Cebula G, Correia VG, Cimpoesu D, Raffay V, Trenkler S, Markota A, Stromsoe A, Burkart R, Perkins GD, Bossaert LL; EuReCa ONE Collaborators. Corrigendum to "EuReCa ONE-27 Nations, ONE Europe, ONE Registry A prospective one month analysis of out-of-hospital cardiac arrest outcomes in 27 countries in Europe" [Resuscitation 105 (2016) 188-195]. Resuscitation. 2016 Dec;109:145-146. doi: 10.1016/j.resuscitation.2016.10.001. Epub 2016 Oct 15. No abstract available. PMID 27750053
- [Background] Kern KB, Hilwig RW, Berg RA, Sanders AB, Ewy GA. Importance of continuous chest compressions during cardiopulmonary resuscitation: improved outcome during a simulated single lay-rescuer scenario. Circulation. 2002 Feb 5;105(5):645-9. doi: 10.1161/hc0502.102963. PMID 11827933
- [Background] Pollack RA, Brown SP, Rea T, Aufderheide T, Barbic D, Buick JE, Christenson J, Idris AH, Jasti J, Kampp M, Kudenchuk P, May S, Muhr M, Nichol G, Ornato JP, Sopko G, Vaillancourt C, Morrison L, Weisfeldt M; ROC Investigators. Impact of Bystander Automated External Defibrillator Use on Survival and Functional Outcomes in Shockable Observed Public Cardiac Arrests. Circulation. 2018 May 15;137(20):2104-2113. doi: 10.1161/CIRCULATIONAHA.117.030700. Epub 2018 Feb 26. PMID 29483086
- [Background] Nolan JP, Soar J, Zideman DA, Biarent D, Bossaert LL, Deakin C, Koster RW, Wyllie J, Bottiger B; ERC Guidelines Writing Group. European Resuscitation Council Guidelines for Resuscitation 2010 Section 1. Executive summary. Resuscitation. 2010 Oct;81(10):1219-76. doi: 10.1016/j.resuscitation.2010.08.021. No abstract available. PMID 20956052
- [Background] Perkins GD, Olasveengen TM, Maconochie I, Soar J, Wyllie J, Greif R, Lockey A, Semeraro F, Van de Voorde P, Lott C, Monsieurs KG, Nolan JP; European Resuscitation Council. European Resuscitation Council Guidelines for Resuscitation: 2017 update. Resuscitation. 2018 Feb;123:43-50. doi: 10.1016/j.resuscitation.2017.12.007. Epub 2017 Dec 9. No abstract available. PMID 29233740
- [Background] Becker TK, Berning AW, Prabhu A, Callaway CW, Guyette FX, Martin-Gill C. An assessment of ventilation and perfusion markers in out-of-hospital cardiac arrest patients receiving mechanical CPR with endotracheal or supraglottic airways. Resuscitation. 2018 Jan;122:61-64. doi: 10.1016/j.resuscitation.2017.11.054. Epub 2017 Nov 23. PMID 29175355
- [Background] Axelsson C, Karlsson T, Axelsson AB, Herlitz J. Mechanical active compression-decompression cardiopulmonary resuscitation (ACD-CPR) versus manual CPR according to pressure of end tidal carbon dioxide (P(ET)CO2) during CPR in out-of-hospital cardiac arrest (OHCA). Resuscitation. 2009 Oct;80(10):1099-103. doi: 10.1016/j.resuscitation.2009.08.006. Epub 2009 Aug 28. PMID 19716640
- See also: Hjärt-lungräddningsregistret årsrapport 2017. Stockholm: HLR rådet — https://hlr.se/